CLINICAL TRIAL: NCT07236151
Title: A Clinical Study of Sequential CD19/CD22 CAR-T Cell Therapy Following Autologous Stem Cell Transplantation in Relapsed/Refractory Large B-cell Lymphoma
Brief Title: Sequential CD19/CD22 CAR-T Cell Therapy Following ASCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASCT+CD19/22 CART
Record Dates: First submitted 2025-09-26; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Large B-cell Lymphoma; CAR T Cell Therapy; Auto Stem Cell Transplant
MeSH Terms: interventions — Blood Component Removal; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASCT+ CD19/CD22 CAR-T (Experimental)
  Interventions: Other: Apheresis and Bridging Therapy; Other: Conditioning and Stem Cell Transplantation; Other: CAR-T Cell Administration

INTERVENTIONS:
Other: Apheresis and Bridging Therapy — Patients undergo two separate apheresis procedures:
  * Mobilization and collection of autologous hematopoietic stem cells (HSCs) .
  * Collection of peripheral blood mononuclear cells (PBMCs) for the manufacture of CD19 and CD22 CAR-T cell products.
  Bridging therapy may be administered at the investigator's discretion between apheresis and the conditioning regimen.
  Other Names: 1
Other: Conditioning and Stem Cell Transplantation — Patients undergo a myeloablative conditioning regimen, followed by the infusion of autologous hematopoietic stem cells on Day 0.
  Other Names: 2
Other: CAR-T Cell Administration — Fractionated infusions of CD19-directed and CD22-directed CAR-T cells are completed within one week after HSC infusion.
  Other Names: 3

SUMMARY:
The goal of this clinical trial is to learn if sequential CD19/CD22 CAR-T cell therapy following autologous stem cell transplantation (ASCT) works to treat relapsed or refractory large B-cell lymphoma (LBCL) in adults. It will also learn about the safety of this treatment combination. The main questions it aims to answer are:

Does ASCT followed by sequential CD19/CD22 CAR-T therapy improve complete response rates in participants with relapsed/refractory LBCL? What medical problems do participants have when receiving this treatment combination? Researchers will evaluate the safety and efficacy of ASCT followed by sequential CD19/CD22 CAR-T therapy to determine if this treatment approach works to improve outcomes for patients with relapsed/refractory LBCL.

Participants will:

Undergo two separate apheresis procedures for stem cell collection and CAR-T cell manufacturing.

Receive conditioning chemotherapy followed by autologous stem cell infusion on day 0.

Receive sequential CD19 and CD22 CAR-T cell infusions over 3 days within one week post-transplant.Visit the clinic regularly for checkups and tests to monitor their response to treatment and any potential side effects.

Keep a record of their symptoms and any adverse events experienced during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed or refractory large B-cell lymphoma (LBCL) after at least one prior line of therapy.

   *[Note: LBCL includes: diffuse large B-cell lymphoma, not otherwise specified (DLBCL-NOS); diffuse large B-cell lymphoma transformed from follicular lymphoma (FL-DLBCL); grade 3b follicular lymphoma (FL); primary mediastinal large B-cell lymphoma (PMBCL); high-grade B-cell lymphoma with rearrangements of MYC and BCL-2 and/or BCL-6 (double-hit/triple-hit lymphoma, DHL/THL)].*
2. Age Restriction: Individuals must be 18 to 70 years old.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
4. Presence of at least one measurable target lesion. *[Note: A target lesion is defined as ≥1 lesion with a longest diameter (LD) >1.5 cm and a longest perpendicular diameter (LPD) ≥1.0 cm, as assessed by computed tomography (CT) or magnetic resonance imaging (MRI).]*
5. Adequate organ function, defined as:

   * Left ventricular ejection fraction (LVEF) ≥50% by echocardiography;
   * Creatinine clearance ≥30 mL/min;
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × upper limit of normal (ULN).
6. Adequate hematopoietic function, defined as:

   * Platelet count ≥45 ×10⁹/L;
   * Hemoglobin ≥8.0 g/dL;
   * Absolute neutrophil count (ANC) ≥1.0 × 10⁹/L.
7. Life expectancy ≥3 months.
8. For women of childbearing potential, a negative pregnancy test is required. Both male and female patients must agree to use effective contraception during treatment and for 1 year thereafter.
9. Willingness to provide written informed consent.

Exclusion Criteria:

1. Prior allogeneic hematopoietic stem cell transplantation or CAR-T cell therapy.
2. Use of immunosuppressive agents or systemic corticosteroids (equivalent to >10 mg prednisone daily) within 2 weeks prior to leukapheresis, or requirement for continued use after enrollment.
3. Active hepatitis B (HBsAg positive with detectable HBV DNA) or hepatitis C (anti-HCV positive with detectable HCV RNA) infection at screening.
4. Uncontrolled active infection requiring intravenous antimicrobial therapy.
5. History of other malignancies within 2 years prior to enrollment (except adequately treated basal cell carcinoma of skin, squamous cell carcinoma of skin, or carcinoma in situ).
6. Significant comorbidities that may compromise study participation or patient safety, including:

   * Severe cardiovascular disease (NYHA Class III/IV heart failure, myocardial infarction within 6 months, unstable arrhythmias, or angina)
   * Severe pulmonary dysfunction (FEV1 or DLCO ≤50% predicted, or requiring supplemental oxygen)
7. HIV infection (positive serology with detectable viral load).
8. Pregnancy, lactation, or unwillingness to use effective contraception.
9. Any condition that in the investigator's judgment would preclude safe participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Best Complete Response Rate | From the date of CAR-T cell infusion until the end of the study, with an average follow-up period of approximately 2 years.
  Best Complete Response Rate (CRR), defined as the proportion of patients achieving a best response of complete response according to the Lugano 2014 criteria.

SECONDARY OUTCOMES:
Overall survival | From the date of CAR-T cell infusion until the date of death or last follow-up, assessed up to 5 years.
Event-free survival | From the date of CAR-T cell infusion to the date of first event (disease progression, relapse, or death) or last follow-up, assessed up to 5 years.
Adverse event | Within 30 days after CAR-T cell infusion
Best Overall Response Rate | From the date of CAR-T cell infusion until the end of the study, with an average follow-up period of approximately 2 years.
  Best Overall Response Rate (ORR), defined as the proportion of patients achieving a best response of complete response (CR) or partial response (PR) according to the Lugano 2014 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No